CLINICAL TRIAL: NCT02524106
Title: Bococizumab HIV Evaluation (B-HIVE) Study: A Phase 3, Double-Blind, Randomized, Placebo-Controlled Study to Assess the Efficacy and Safety of Bococizumab, a PCSK9 Inhibitor, in HIV-Infected Subjects
Brief Title: Bococizumab HIV Evaluation (B-HIVE) Study
Acronym: B-HIVE
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Industry won't be moving forward with production of bococizumab
Sponsor: University of California, San Francisco (Other)
Collaborators: Pfizer (Industry); San Francisco General Hospital (Other)
Responsible Party: Principal Investigator, Priscilla Hsue, MD, Principal Investigator, University of California, San Francisco
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: WI204426
Record Dates: First submitted 2015-08-12; First posted 2015-08-14 (Estimated); Results first posted 2019-06-19 (Actual); Last update posted 2019-06-19 (Actual); Status verified 2019-06

CONDITIONS: Dyslipidemia; Cardiovascular Disease
MeSH Terms: conditions — Dyslipidemias; Cardiovascular Diseases | interventions — bococizumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Bococizumab (Experimental): 150 mg bococizumab injected subcutaneously every 2 weeks for a duration of 52 weeks
  Interventions: Drug: Bococizumab
- Placebo (Placebo Comparator): 150 mg placebo injected subcutaneously every 2 weeks for a duration of 52 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Bococizumab — PF-04950615 is a humanized monoclonal antibody against the proprotein convertase subtilisin kexin type 9 (PCSK9) enzyme responsible for the degradation of the low-density lipoprotein receptor (LDLR), being developed by Pfizer, Inc for the treatment of primary hyperlipidemia and mixed dyslipidemia.
  Other Names: PF-04950615
  Arms: Bococizumab
Drug: Placebo — placebo
  Arms: Placebo

SUMMARY:
B-HIVE is a Phase 3, double blind, placebo-controlled, randomized, parallel group study, designed to compare the efficacy and safety of bococizumab 150 mg subcutaneously every 2 weeks to bococizumab placebo subcutaneously every 2 weeks for LDL-C lowering in HIV-infected subjects.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) due to atherosclerosis continues to be the leading single cause of death in industrialized countries. High serum lipid levels, and especially high low-density lipoprotein cholesterol (LDL-C) levels, have been demonstrated to strongly and directly correlate with CVD risks by numerous epidemiological studies. Moreover, large prospective clinical outcome trials have demonstrated that lowering LDL-C decreases cardiovascular morbidity and mortality (1). A meta-analysis of 26 randomized clinical trials comprising 170,000 participants showed that more intensive statin therapy compared to less intensive regimens will reduce coronary deaths or myocardial infarction by an additional 13% (2).

HIV-infected individuals represent a unique and increasing subset of atherosclerosis. With the advent of antiretroviral therapy, HIV-infected individuals now have much improved survival and are faced with health issues related to aging, including cardiovascular disease. Individuals with HIV have higher rates of coronary events compared to controls even in the setting of treated and suppressed disease and a growing body of literature suggests that they are at increased risk for myocardial infarction, atherosclerosis, and sudden cardiac death (3-5). Many facets of atherosclerosis differ in HIV-infected individuals compared to uninfected individuals with atherosclerosis. HIV-infected patients with acute coronary syndromes are younger and more likely to be males and smokers, with low high density lipoprotein-cholesterol (HDL-C), compared to other acute coronary syndrome patients (6). With respect to pathophysiology, viral replication, antiretroviral drugs and inflammation all contribute to atherosclerosis (7,8).

HIV-associated inflammation induces pro-atherogenic lipid abnormalities and anti-retroviral therapy leads to the development of metabolic abnormalities such as dyslipidemia, lipodystrophy and insulin resistance (9,10) In a large cross-sectional study, 27% of subjects receiving combination therapy including a protease inhibitor had a total cholesterol level exceeding 240 mg/dl, compared to 8% of untreated HIV subjects, and 40% had triglyceride levels above 200 mg/dl, compared to 15% in untreated subjects (11). The prevalence and severity of dyslipidemia varies among different antiretroviral drugs; (9) however, hypertriglyceridemia and low HDL-cholesterol were associated with HIV infection even before the advent of antiretroviral therapy (12). Total, HDL-C, and LDL-C decrease at the time of HIV infection, and with antiretroviral treatment total and LDL-C levels increase to pre-infection levels while HDL-C remains low (13).

Abnormalities in body composition have been reported in 40-50% of HIV-infected patients, with higher rates in those receiving combination antiretroviral therapy (9). Subcutaneous lipoatrophy commonly affects the face, limbs, and buttocks, and is accompanied by central fat accumulation. Hyperinsulinemia is often also present. In a representative study, (14) diabetes was present in 7% of HIV-infected adults with fat accumulation or lipoatrophy, as compared to 0.5% of control subjects matched for age and BMI. The corresponding rates of glucose intolerance were 35% and 5% respectively (14). Compared to healthy control subjects, HIV-infected men treated with combination antiretroviral therapy were 4 times as likely to develop diabetes over a 3-year observation period (15).

The increased cardiovascular risk and dyslipidemia in HIV-infected individuals is difficult to treat for several reasons. Statins reduce LDL-C levels less in HIV-infected individuals compared to uninfected controls (16). Fibrates reduce triglyceride levels less in HIV-infected individuals compared to uninfected controls as well (16). Drug-drug interactions between statins and protease inhibitors increase the risk of adverse events (17,18). Due to these interactions, simvastatin and lovastatin are contraindicated among individuals receiving protease inhibitors and the dose of atorvastatin should not exceed 40 mg (17). Even interactions with rosuvastatin, which is not metabolized by the cytochrome P450 system, have been described (19,20).

As a consequence, physicians may avoid treating HIV-infected individuals who would benefit from statins, or use lower doses or less potent statins, reducing the potential for cardiovascular event reduction. High triglyceride levels in HIV-infected subjects are common, and the combination of a fibrate plus antiretroviral therapy increases the risk of drug-drug adverse events, even before consideration of a statin.

Statin treatment reduces lipid levels modestly in HIV subjects. Among 72 HIV-infected subjects in the SATURN-HIV trial randomized to rosuvastatin 10 mg/day, LDL-C was reduced by 25.3% by week 24 (21). In another study, of 83 HIV-infected subjects, rosuvastatin 10 mg and pravastatin 40 mg/day reduced LDL-C by 37% and 19% respectively at 45 days (22). Among 151 HIV-infected subjects randomized to rosuvastatin 10 mg, atorvastatin 10 mg, or pravastatin 40 mg/day, LDL-C reductions were greater with rosuvastatin at this dose, but all 3 statins significantly and similarly reduced serum levels of hs-CRP and TNF (23).

That statins might favorably influence the evolution of atherosclerosis in HIV-infected subjects is suggested by a recent trial where 40 HIV subjects with mild coronary atherosclerosis by CT angiography and aortic inflammation by FDG-PET imaging were randomized to atorvastatin 20-40 mg/day or placebo and were followed for 12 months (24). Atorvastatin significantly reduced non-calcified coronary plaque volume relative to placebo, as well as the number of high-risk plaques.

Approximately 1/3 of individuals with HIV-infection are co-infected with hepatitis C (25). Elevated hepatic enzymes due to hepatitis C represent a relative contraindication to statin therapy, and some evidence suggests that a statin might increase hepatitis C activity (26). Finally, HIV-infected patients often need many medications and have a large daily pill burden. Compliance suffers, but has been shown to improve when single tablet regimens reduce daily pill load.27 Long-acting injectable antiretroviral drugs are under development as a strategy to reduce pill burden and improve compliance (28). PCSK9 inhibitor injections would dovetail well with this approach. For these reasons, PCSK9 inhibitor therapy offers advantages over statin therapy in this unique population.

Bococizumab (RN316/PF-04950615) is a novel humanized PCSK9 monoclonal antibody. In a 24-week, multicenter, randomized, double-blind, placebo-controlled phase II trial, the LDL-C lowering effects of bococizumab, administered every 2 or 4 weeks in statin-treated adults with LDL-C ≥80 mg/dL was assessed (29). Subjects were randomized to placebo, bococizumab 50 mg, 100 mg, or 150 mg every 2 weeks, or placebo, bococizumab 200 mg or 300 mg monthly. The dose was reduced if LDL-C was ≤25 mg/dL. The primary analysis was the placebo-adjusted treatment difference for the change from baseline in LDL-C at week 12.

Overall, 354 patients were randomized, 351 received study treatment, and 299 completed the study. Bococizumab significantly reduced LDL-C across all doses. The placebo-adjusted LDL-C reduction at 12 weeks for the 2-weekly dosing regimen was 34.3% with 50 mg, 45.1% for 100 mg and 53.4% for 150 mg, and for the monthly dosing regimen was 27.6% for 200 mg and 44.9% for 300 mg. The incidence and profile of adverse events were similar across placebo and bococizumab groups.

Based on these findings, 150 mg every 2 weeks was selected as the dose for phase III trials, including this trial. Because multiple doses of bococizumab as high as 150 mg every 2 weeks and 300 mg every 4 weeks up to 12 weeks were safe and well tolerated, the primary rationale for dose selection was the pharmacokinetic/pharmacodynamic model that predicted LDL-C change from baseline. Based on population PK/PD modeling, a dose of 150 mg every 2 weeks in patients on a background of statins is estimated to be equivalent to approximately 80% of the maximal response for LDL-C lowering (-67%). Assuming an average LDL C at baseline of 100 mg/dL for HIV-infected individuals, the mean absolute LDL-C reduction is predicted to be approximately 60 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

1. Evidence of a personally signed and dated informed consent document indicating that the subject (or a legal representative) has been informed of all pertinent aspects of the study.
2. Subjects who are willing and able to comply with scheduled visits, treatment plan, laboratory tests, and other study procedures.
3. Males and females greater than 40 years of age.
4. With documented HIV infection.
5. Moderate or high CVD risk defined as:

   documented CVD as assessed by meeting at least 1 of 3 criteria below:
   1. Coronary artery disease (CAD): prior MI due to atherosclerosis, coronary artery bypass graft surgery, percutaneous coronary intervention, or angiographic CAD with luminal diameter stenosis of at least one coronary artery at least 50%.
   2. Cerebrovascular disease: prior ischemic stroke of carotid origin, carotid endarterectomy or stenting, or angiographic carotid stenosis of at least 50%.
   3. Peripheral arterial disease: prior lower extremity arterial surgical or percutaneous revascularization procedure, or angiographic lower extremity arterial stenosis of at least 50%.

   OR any one of the following CVD risk factors:
   1. Controlled type II diabetes mellitus (HbA1C ≤8.0% within the past 90 days prior to study entry, regardless of use of medications)
   2. Current smoking: participant report of smoking at least a half a pack of cigarettes a day, on average, in the past month.
   3. Hypertension: two consecutive BP readings with either systolic >140 mmHg or diastolic >90 mmHg; or on antihypertensive medications.
   4. Dyslipidemia: defined as or HDL-C ≤ 40 mg/dL for men or ≤50 mg/dL for women, regardless of medication use.
   5. a hsCRP ≥2mg/L at screening.
6. Lipids at screening visit:

   * Fasting LDL-C 70 mg/dL (1.81 mmol/L);
   * Fasting TG ≤ 600 mg/dL (6.78 mmol/L).
7. Male and female subjects of childbearing potential must agree to use a highly effective method of contraception throughout the study and for at least 63 days after the last dose of assigned treatment. A subject is of childbearing potential if, in the opinion of the investigator, he/she is biologically capable of having children and is sexually active.

Female subjects who are not of childbearing potential (ie, meet at least one of the following criteria):

* Have undergone a documented hysterectomy or bilateral oophorectomy;
* Have medically confirmed ovarian failure; or
* Achieved post menopausal status, defined as: cessation of regular menses for at least 12 consecutive months with no alternative pathological or physiological cause; and have a serum follicle stimulating hormone (FSH) level within the laboratory's reference range for postmenopausal females.

Exclusion Criteria:

1. Subjects who are investigational site staff members directly involved in the conduct of the trial and their family members, site staff members otherwise supervised by the Investigator, or subjects who are Pfizer employees.
2. Participation in other studies involving small molecule investigational drug(s) (Phases 1 4) within 1 month 5 half lives, whichever is longer except for cholesteryl ester transfer protein (CETP) inhibitors (indefinitely), or biological agents within 6 months or 5 half lives, whichever is longer before the current study begins and/or during study participation (the investigator should refer to documents provided by the subject on the other study to determine the investigational product half life). If the blind has been broken and the Investigator knows (with documentation) that the subject received placebo, he/she can be included.
3. Subjects with prior exposure to bococizumab or another PCSK9 inhibitor.
4. Subjects who are unable to receive injections, as either a self-injection, or administered by another person.
5. History of a cardiovascular or cerebrovascular event or procedure (eg, myocardial infarction, stroke, transient ischemic attack, angioplasty) during the past 90 days.
6. Congestive heart failure, New York Heart Association functional class IV, or left ventricular ejection fraction measured by imaging known to be <25%. (Imaging not required for study inclusion).
7. Poorly controlled hypertension (on or off treatment) at screening visit or at randomization (defined as the average of two systolic blood pressure (BP) measurements greater than 160 mm Hg or the average of two diastolic BP measurements greater than 100 mm Hg).
8. Any history of hemorrhagic stroke or lacunar infarct.
9. CD4 count at screening visit <350 cells/mm3.
10. Current untreated hypothyroidism or thyroid stimulating hormone (TSH) >1 X upper limit of normal (ULN) at screening. Subjects who are treated and well controlled should be on a stable dose of thyroid hormone for at least 6 months.
11. Current history of alcoholism or drug addiction according to the Diagnostic and Statistical Manual of Mental Disorders (DSM) IV criteria within 12 months prior to screening. Use of any recreational drugs within 12 months prior to screening.
12. History of cancer within the last 5 years (except for cutaneous basal cell or squamous cell cancer resolved by excision, or cervical carcinoma in si tu).
13. Any disease or condition that might compromise the hematological, renal, hepatic, pulmonary, endocrine, central nervous, immune, or gastrointestinal systems (unless deemed not clinically significant by the Investigator and/or the Sponsor) or confound the interpretation of the study results. Examples of such conditions include but are not limited to nephrotic syndrome, uncontrolled diabetes, excessive alcohol consumption, cholestatic liver disease, unstable mental illness.
14. Undergoing apheresis or have a planned start of apheresis.
15. Initiation of or change in non-lipid lowering prescription drugs, herbal medicine or supplements (including foods with added plant sterols and stanols) within 6 weeks of screening with the exception of initiation or change in multivitamins used for general health purposes. Short-term use of medications to treat acute conditions, and vaccines are allowed (e.g., antibiotics or allergy medication).
16. History of allergic or anaphylactic reaction to any therapeutic or diagnostic monoclonal antibody (IgG protein) or molecules made of components of monoclonal antibodies (eg, Enbrel® which contains the Fc portion of an antibody or Lucentis® which is a Fab).
17. Any abnormal hematology values, clinical chemistries, or ECGs at screening judged by the Investigator as clinically significant, which could impact on subject safety, were the potential subject to be included in the study, or interfere with the interpretation of study results.
18. Active phase hepatitis. Stable patients with hepatitis B or C infection >2 years before randomization are eligible.
19. Aspartate transaminase (AST) or alanine transaminase (ALT) >5 X ULN at screening.
20. Direct bilirubin >4.0 X ULN at screening.
21. GFR <30 mL/min/1.73m2 at screening or undergoing dialysis.
22. Plans to donate blood during the study.
23. Pregnant females; breastfeeding females.
24. Additional exclusion criteria for the FDG-PET/CT imaging (patients with these exclusions may participate in the rest of the trial):

    1. Significant radiation exposure during the year prior to randomization. Significant exposure is defined as i) more than 2 PCI procedures, ii) more than 2 myocardial perfusion studies, or iii) more than 2 CT angiograms.
    2. Any history of radiation therapy.
    3. Current insulin use.
25. Additional exclusion criteria for CTA imaging (patients with these exclusions may participate in the rest of the trial):

    1. Significant radiation exposure during the year prior to randomization. Significant exposure is defined as i) more than 2 PCI procedures, ii) more than 2 myocardial perfusion studies, or iii) more than 2 CT angiograms (as with FDG-PET/CT.
    2. Any history of radiation therapy (as with FDG-PET/CT).
    3. Any contraindication to beta-blocker or nitroglycerin use, because these drugs are given as part of the standard cardiac CT protocol.
    4. Significant renal dysfunction (defined as an eGFR <60 mL/min/1.73m2).
    5. Body weight >300 pounds (136 Kg), because of the CT scanner table limitations.
    6. Allergy to iodine-containing contrast media.

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2016-08; Primary Completion 2017-11 (Actual); Study Completion 2017-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Priscilla Y Hsue, MD, Principal Investigator — priscilla.hsue@ucsf.edu
Locations (3):
- United States (3):
  - San Francisco General Hospital, San Francisco, California
  - Quest Clinical Research, San Francisco, California
  - San Francisco Veteran's Affair Medical Center, San Francisco, California

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Bococizumab | Placebo
Started | 6 | 5
Completed | 6 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Bococizumab | Placebo | Total
Number analyzed (Participants) | 6 | 5 | 11
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 2 | 3 | 5
  >=65 years | 4 | 2 | 6
Age, Continuous [Mean (Full Range); unit: years] | 64.83 [48 to 73] | 55.4 [40 to 67] | 56.5 [40 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 1 | 1
  Male | 6 | 4 | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: Caucasian | 2 | 2 | 4
  Race/Ethnicity: African-American | 3 | 2 | 5
  Race/Ethnicity: Hispanic | 1 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 6 | 5 | 11
Absolute CD4 T cell [Mean (Full Range); unit: cells/mm3] | 427 [163 to 438] | 834.8 [510 to 1203] | 612.4 [163 to 1203]

OUTCOME MEASURES:

1. Primary Outcome: Change of LDL-C From Baseline to Week 12
Description: The primary endpoint for the study is the percent change from baseline in fasting LDL-C at week 12.
Time Frame: week 12
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Bococizumab | Placebo
Number analyzed (Participants) | 6 | 5
percentage change | 115.3 [75 to 170] | 90.3 [61 to 107]
Statistical Analysis 1: Comparison: Bococizumab vs Placebo; Test type: Other; p = 0.028, Mixed Models Analysis; percentage difference = 61

2. Secondary Outcome: Change in Lp(a) From Entry to Week 12
Description: The primary endpoint for the study is the percent change from baseline in fasting total Lp(a) at week 12.
Time Frame: week 12
Population: Patients living with well controlled HIV
Measure: Mean (Full Range); unit: percentage change
Arm/Group | Bococizumab | Placebo
Number analyzed (Participants) | 6 | 5
percentage change | 327863.05 [54502.5 to 601223.6] | 344580.15 [49758.5 to 639401.8]
Statistical Analysis 1: Comparison: Bococizumab vs Placebo; Test type: Other; p = 0.096, Mixed Models Analysis; percentage difference = 39

ADVERSE EVENTS:
Time Frame: 9 months
Arm/Group | Bococizumab | Placebo
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/5
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/5
Other Adverse Events (participants affected / at risk) | 0/6 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-10): https://cdn.clinicaltrials.gov/large-docs/06/NCT02524106/Prot_SAP_000.pdf